CLINICAL TRIAL: NCT01546805
Title: The Effect of Zinc Supplementation on the Efficacy and Duration of Botulinum Toxin for the Treatment of Oculofacial Spasm Disorders
Brief Title: Testing the Effect of Zinc Supplementation to Improve the Treatment Effect of Botulinum Toxin for Oculofacial Spasm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R.P. #11-3601
Record Dates: First submitted 2012-02-16; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Blepharospasm; Hemifacial Spasm
Keywords: Blepharospasm; Hemifacial spasm; Botox; Zinc
MeSH Terms: conditions — Blepharospasm; Hemifacial Spasm | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Sugar pill
- Zinc Group (Experimental)
  Interventions: Drug: Zinc Supplement

INTERVENTIONS:
Drug: Zinc Supplement — The interventional group will be requested to take zinc supplements (50mg), once daily starting 5 days prior to Botox injections and to be continued for 5 days after injection.
  Arms: Zinc Group
Drug: Sugar pill — The control group will be requested to take placebo pills, once daily starting 5 days prior to Botox injections and to be continued for 5 days after injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether zinc supplements are effective in enhancing the treatment of oculofacial spasm disorders with botulinum toxin.

DETAILED DESCRIPTION:
Botulinum Toxin (Botox) has been used for many years in the treatment of oculofacial dystonias such as blepharospasm and hemifacial spasm. It has also gained widespread use for cosmetic purposes. The efficacy and duration of its effect is not constant amongst all patients. Some patient respond very well, while others have no clinical benefit or the clinical benefit does not last as long as expected. Zinc is known to be an important co-factor in the molecular effects of Botox. The investigators hypothesize that one of the many factors that may contribute to the variability in the response to Botox may be the level of Zinc available within the neuromuscular junction of those patients. The investigators plan to to test whether or not giving patients supplemental Zinc with their Botox injections would help improve the magnitude and duration of the intended clinical effect.

ELIGIBILITY:
Inclusion Criteria:

* greater than the age 18 years old
* patient with hemifacial spasm
* patient with benign essential blepharospasm.

Exclusion Criteria:

* patients who have received Botox within 3 months time,
* patients prone to malabsorption (i.e. those with Celiac disease, inflammatory bowel disease, liver disease, laxative use)
* patients who cannot tolerate zinc supplementation due to kidney disease, gastrointestinal disease, or any other medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Jankovic Rating Scale | 3 months post Botox injection
  a well established scale used in the literature to grade the symptoms of patients with facial spasms disorders.

SECONDARY OUTCOMES:
Treatment Duration Cycle | The time frame will vary with each patient. The time frame is in fact the outcome measure being measured. On average the Botox treatment cycles last 3 months, however this average may be affected by zinc supplements.
  The number of days between the date of Botox injection to the date in which the symptoms have returned back to baseline.
Blepharospasm Disability Index (BDI) | 3 months post Botox injection
  BDI is a scale commonly used in the Blepharospasm literature to measure the magnitude of the burden of symptoms in patients with Blepharospasm. It has also been used to measure treatment effect by a reduction in patient's BDI.

CONTACTS AND LOCATIONS:
Overall Officials: John Harvey, MD, Principal Investigator — St Joseph's Hospital Hamilton; Yasser Khan, MD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - St Joseph's Hospital Hamilton, Hamilton, Ontario
  - Carrot Eye Centre, Mississauga, Ontario